CLINICAL TRIAL: NCT01747317
Title: Individual-Patient-Data Pooled-Analysis of Diagnostic Accuracy of Noninvasive Fractional Flow Reserve From Anatomic CT Angiography
Brief Title: Diagnostic Performance of Noninvasive Fractional Flow Reserve From Computed Tomography
Acronym: PERFECT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, MD,FACC, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TENTH1010
Record Dates: First submitted 2012-12-09; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease
Keywords: FFR; fractional flow reserve; CT; Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Experimental): Single arm study.The investigators will conduct computed tomography,angiography and FFR measurement during angiography in this single arm.
  Interventions: Device: FFR (PressureWire)

INTERVENTIONS:
Device: FFR (PressureWire) — Fractional flow reserve measured during cardiac catheterization--A pressure-monitoring guidewire(PressureWire Certus, St. Jude Medical Systems, Uppsala, Sweden;ComboWire, Volcano Corporation, San Diego, California) will be advanced past the stenosis.
  Other Names: PressureWire™ Certus(St. Jude Medical Systems); PressureWire™ Certus(ComboWire, Volcano Corporation)

SUMMARY:
Fractional Flow Reserve derived from computed tomography(FFRCT) is a novel method for determining the physiologic significance of coronary artery disease (CAD), which will help physicians in clinical decision-making and decrease the medical cost, but its ability to identify patients with ischemia has not been adequately examined to date.

DETAILED DESCRIPTION:
Fractional Flow Reserve derived from computed tomography(FFRCT) is a novel method for determining the physiologic significance of coronary artery disease (CAD), which will help physicians in clinical decision-making and decrease the medical cost, but its ability to identify patients with ischemia has not been adequately examined to date.

Available data from registered clinical trials has testified the diagnostic performance of FFRCT, but the diagnostic accuracy among them are not consistent.

Thus, the investigators designed a collaborative individual patient-data pooled-analysis aimed to assess the diagnostic accuracy of FFRCT and find the possible cause for inconsistency

ELIGIBILITY:
Inclusion Criteria:

* Coronary computed tomographic angiography(CCTA) with over 50 percent stenosis in a major coronary artery over 2mm diameter
* Undergoing clinically indicated invasive coronary angiography with FFR

Exclusion Criteria:

* A history of CABG surgery
* Prior percutaneous coronary intervention with suspected instent restenosis
* Suspicion of or recent acute coronary syndrome
* Complex congenital heart disease
* Prior pacemaker or defibrillator
* Prosthetic heart valve
* Significant arrhythmia
* heart rate >100 beats/min
* systolic blood pressure≤90 mmHg
* contraindication to beta blockers, nitroglycerin or adenosine
* Serum creatinine level greater than 1.5 mg per dL
* Allergy to iodinated contrast
* Pregnant state
* Body mass index greater than 35
* Evidence of active clinical instability or lifethreatening disease
* Canadian Cardiovascular Society class IV angina
* nonevaluable CCTA as determined by the CCTA core laboratory
* Inability to adhere to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of FFRCT | 1 day
  Diagnostic accuracy[Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV)]* of FFRCT to determine presence or absence of at least one hemodynamically (HD)-significant coronary artery stenosis at the subject level using binary outcomes when compared to FFR as the reference standard..*Sensitivity measures the proportion of actual positives which are correctly identified. Specificity measures the proportion of negatives which are correctly identified;PPV, or precision rate is the proportion of positive test results that are true positives (such as correct diagnoses);NPV is defined as the proportion of subjects with a negative test result who are correctly diagnosed.

SECONDARY OUTCOMES:
Diagnostic accuracy of FFRCT at the subject level | 1 day
  Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of FFRCT at the subject level using binary outcomes when compared to FFR as the reference standard.
Diagnostic accuracy of FFRCT at the vessel level | 1 day
  Sensitivity, specificity, PPV and NPV of FFRCT for the presence or absence of HD-significant coronary artery stenosis at the vessel level using binary outcomes when compared to FFR as the reference standard.
FFR Numerical Correlation | 1 day
  Per-vessel correlation of the FFRCT numerical value alone with the FFR numerical value measured during cardiac catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Wei Xu, MD, FACC, Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital, Tongji University School of Medicine
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, China

REFERENCES:
- [Result] Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J, Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. J Am Coll Cardiol. 2011 Nov 1;58(19):1989-97. doi: 10.1016/j.jacc.2011.06.066. PMID 22032711
- [Result] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562